CLINICAL TRIAL: NCT04209491
Title: "Pilot Study: Interest of the Intervention of a Nurse Coordinator in Complex Care Pathway in the Management of a Patient Treated for Hepatocellular Carcinoma (HCC)"
Brief Title: Interest of the Intervention of a Nurse Coordinator in Complex Care Pathway
Acronym: INFIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 180129
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is based on the assumption that the nurse coordinators of the centres have common missions at each of the key stages of patient care. These missions make the care plan more fluid and improve the quality and safety of care as well as the patient's prognosis.

The Hypothesis is that co-follow-up by a doctor and a nurse coordinator reduces time between referral to treatment, average lengths of stay, unscheduled readmissions or early emergency visits, compared to follow-up that does not involve a nurse coordinator.

DETAILED DESCRIPTION:
Main objective:

Describe the roles and missions of professionals dedicated to the coordination of care pathways for patients with HCC

Secondary objectives:

Compare the indicators of quality of care in HCC centres with a nurse coordinator:

1. Timeframe in treatment:

   * timeframe between the first contact with the HCC centre and the first interventional radiology treatment.
   * timeframe between the first contact with the centre and the first presentation at a multidisciplinary team meeting (MDT)
   * time between the first contact with the centre and the diagnostic consultation
   * timeframe between the first contact with the centre and discharge from the hospital
   * timeframe between the first interventional radiology procedure and the next for the subgroup of patients who have multiple procedures during the follow-up period
   * timeframe between the first contact with the nurse coordinator of the centre and discharge from the hospital.
2. The average length of stay of hospitalization
3. The number of visits to the emergency unit during the first month following the radiology intervention
4. The number of unscheduled readmissions during the first month following the intervention.

Assess the feasibility of collecting the above-mentioned timeframe and variables and the patients and carers feedback on the coordination of the care pathway Describe the organization of care pathways for patients with HCC in centres with or without a nurse coordinator.

Research method: This is a retrospective descriptive pilot study. It aims to describe the organization of care.

Population: Patient with a diagnosis of localized hepatocellular carcinoma.

Data processing:

* Feasibility questionnaires will be sent by email.
* The interviews will be transcribed and coded with NVivo® software
* Patient data will be collected in the ecrf
* Data processing from anonymized files by the authors of the research only. All data will be centralized at Bichat Hospital (URC Paris Nord) for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Centre with interventional radiology treatment
* Active list of patients followed for a HCC of at least 70 / year
* Reply to the feasibility questionnaire within 60 days from receipt of the email

Exclusion Criteria:

* Patient with a localized HCC diagnosis (BCLC A or B)
* Hospitalised for a first interventional radiology treatment (radioembolisation, transarterial chemoembolization or percutaneous ablation) in one of the centres included in the study between July 1, 2017 and December 31, 2017

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a diagnosis of localized hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of the following missions of the coordinator Nurse | 12 months
  missions: o Initial contact of the patient with the expert centre
  * Organisation of the MDT meeting
  * Organisation of treatment and investigations
  * Coordination between hospital professionals
  * Link with community health professionals
  * Follow-up (post-hospitalization, treatment side effects, etc.)
  * Information, advice to patients
  * Psychological support
  * Implementation of care pathways
  * Nursing research

SECONDARY OUTCOMES:
Timeframe in days between The first contact with the centre and the first interventional radiology treatment. | 12 months
  Timeframe in days between The first contact with the centre and the first interventional radiology treatment.
Timeframe in days between : The first contact with the centre and the first presentation at a MDT meeting | 12 months
  Timeframe in days between : The first contact with the centre and the first presentation at a MDT meeting
Timeframe in days between : The first contact with the centre and the diagnostic consultation | 12 months
  Timeframe in days between : The first contact with the centre and the diagnostic consultation
Timeframe in days between :The first contact with the centre and discharge from the hospital | 12 months
  Timeframe in days between :The first contact with the centre and discharge from the hospital
Timeframe in days between :The interventional radiology procedure and the next one for the subgroup of patients who have multiple procedures during the follow-up period | 12 months
  Timeframe in days between :The interventional radiology procedure and the next one for the subgroup of patients who have multiple procedures during the follow-up period
Length of hospital stay for a first interventional radiology treatment in patients with HCC. | 12 months
  Length of hospital stay for a first interventional radiology treatment in patients with HCC.
Number of emergency unit visits during the first month following hospitalization for interventional radiology treatment for patients included in the study. | 12 months
  Number of emergency unit visits during the first month following hospitalization for interventional radiology treatment for patients included in the study.
Number of early unscheduled readmissions during the first month following interventional radiology treatment for patients included in the study. | 12 months
  Number of early unscheduled readmissions during the first month following interventional radiology treatment for patients included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Julie DEVICTOR, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- BEAUJON Hospital, Clichy-sous-Bois, France